CLINICAL TRIAL: NCT01222728
Title: Using Positron Emission Tomography (PET) to Predict Intracranial Tumor Growth in Neurofibromatosis Type II (NF2) Patients
Brief Title: Using Positron Emission Tomography to Predict Intracranial Tumor Growth in Neurofibromatosis Type II Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100193; 10-N-0193
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-06-03

CONDITIONS: Neoplasms; Nervous System Disease; Vestibular Disease
Keywords: PET Imaging; Vestibular Schwannoma; Neurofibromatosis; Neurofibromatosis Type 2; NF2
MeSH Terms: conditions — Neoplasms; Nervous System Diseases; Vestibular Diseases; Neuroma, Acoustic; Neurofibromatoses; Neurofibromatosis 2

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Neurofibromatosis type II (NF2) is associated with tumors of the nerves, brain, and spinal cord. Most people with NF2 develop vestibular schwannomas, or tumors on the hearing and balance nerves. As they grow, vestibular schwannomas can cause hearing loss and balance problems. If they grow very large they can cause more serious problems, such as seizures, loss of eyesight, weakness, speech problems, and problems with the sense of touch. More research is needed into NF2 because researchers do not completely understand why these tumors occur or what makes them grow over time.
* Currently, tumor size is measured with magnetic resonance imaging (MRI) scans. However, MRI scans cannot predict how fast a tumor will grow. By using positron emission tomography (PET) scanning, researchers hope to be able to predict sudden growth spurts of tumors associated with NF2 and develop better treatment methods for this type of cancer.

Objectives:

- To use magnetic resonance imaging and positron emission tomography to better understand the growth of brain tumors in people with neurofibromatosis type II.

Eligibility:

- Individuals between 18 and 50 years of age who have been diagnosed with NF2 and have at least three untreated intracranial tumors.

Design:

* This study requires an initial set of outpatient visits to the NIH Clinical Center that will last 7 to 10 days.
* Participants will have a physical and neurological examination and blood tests at the first visit. Participants will then have the following imaging studies to examine the tumors:
* MRI scans of the brain
* PET scans of the brain, combined with a computed tomography (CT) scan. The PET scans will be performed on separate days. Different contrast agents will be used for both scans, so researchers will inform participants if they need to fast or follow other procedures before having the scan.
* After the initial imaging studies, participants will have additional MRI scans every 6 months for 2 years to track tumor growth.

DETAILED DESCRIPTION:
OBJECTIVE:

The objective of this prospective observational study of intracranial tumors in patients with neurofibromatosis type 2 (NF2) is to gain insight into the use of 18F-fluoro-deoxyglucose (FDG) and 3 -deoxy-3 -18F-fluorothymidine (FLT) positron emission tomography (PET)/computed tomography (CT) as a predictive measure of future tumor growth patterns.

STUDY POPULATION: <TAB>

Twelve patients, ages 18-50, with a clinical or genetic diagnosis of NF2 and harboring at least 3 unoperated intracranial tumors (meningiomas and/or vestibular schwannomas) will participate in this study.

DESIGN:

Study participants will be evaluated with a thorough physical and neurologic examination upon enrollment. This initial outpatient evaluation will include contrast-enhanced magnetic resonance imaging (MRI) of the brain, FDG-PET/CT and FLT-PET/CT scans.

Subjects will be followed as outpatients for two years, during which time MRI evaluation will be performed every six months.

OUTCOME MEASURES:

Based on data derived from this study, we hope to correlate FDG-PET/CT and FLT-PET/CT scans with metabolic activity and cellular proliferation within tumors. These findings will help us better forecast tumor growth and senescence. These findings should permit the safer treatment of the subset of tumors that will grow and cause symptoms and avoid the unnecessary treatment of lesions that will remain stable (not requiring treatment) in these patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Clinical diagnosis of NF2 by established clinical criteria or genetic testing.
* Age 18 to 50.
* A minimum of 3 intracranial tumors (meningiomas and/or VSs) measuring = or > 1cm in size, including:

  1. At least one unoperated VS > 1 cm in size AND
  2. At least one unoperated meningioma > 1 cm in size
* No pregnancy or intent to become pregnant, with proper use of contraception for the duration of the study.
* Normal liver enzymes: tests should be completed within 14 days before injection of the radiopharmaceutical; SGOT, SGPT <5x ULN; bilirubin less than or equal to 2x ULN
* If prior radiation therapy to the tumor: >2 years must have passed after radiotherapy administration and tumor must demonstrate growth after radiotherapy (signifying a viable tumor for study is present)
* If prior chemotherapy: must have completed chemotherapy >6 months prior to enrollment to allow washout of chemotherapeutic agent

EXCLUSION CRITERIA:

* Clinically unstable condition that precludes serial clinical and imaging evaluation (i.e. Class 3 congestive heart failure, severe chronic renal insufficiency, severe chronic obstructive pulmonary disease).
* Contraindication to MRI scanning, including pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, or shrapnel fragments
* Severe chronic renal insufficiency (glomerular filtration rate < 30 mL/min/1.73 m2), hepatorenal syndrome or post-liver transplantation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2010-09-22; Study Completion 2015-06-03

PRIMARY OUTCOMES:
To determine whether FDG and/or FLT uptake correlate with growth rate of meningiomas and Vestibular Schwannomas (VSs) in NF2 patients, and can be used to predict their future growth pattern.

SECONDARY OUTCOMES:
To characterize glucose metabolism and cellular proliferative activity in meningiomas and VSs in NF2 patients, using FDG and FLT PET/CT imaging. To determine the degree to which glucose metabolism and cell proliferation are coupled in meningioma...

CONTACTS AND LOCATIONS:
Overall Officials: John D Heiss, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chen JM, Houle S, Ang LC, Commins D, Allan K, Nedzelski J, Rowed D. A study of vestibular schwannomas using positron emission tomography and monoclonal antibody Ki-67. Am J Otol. 1998 Nov;19(6):840-5. PMID 9831165
- [Background] Abaza MM, Makariou E, Armstrong M, Lalwani AK. Growth rate characteristics of acoustic neuromas associated with neurofibromatosis type 2. Laryngoscope. 1996 Jun;106(6):694-9. doi: 10.1097/00005537-199606000-00007. PMID 8656953
- [Background] Baser ME, Makariou EV, Parry DM. Predictors of vestibular schwannoma growth in patients with neurofibromatosis Type 2. J Neurosurg. 2002 Feb;96(2):217-22. doi: 10.3171/jns.2002.96.2.0217. PMID 11838793